CLINICAL TRIAL: NCT01662583
Title: Pragmatic Clinical Trial of Vaccine Health Literacy Related Text Message Reminders to Increase Receipt of Second Dose of Influenza Vaccine for Young, Low Income, Urban Children
Brief Title: Vaccine Health Literacy Related Text Message Reminders to Increase Receipt of Second Dose of Influenza Vaccine for Young, Low Income, Urban Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAJ9354
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Influenza
Keywords: Influenza; text message; vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Educational Text Message (Experimental): Educational text message reminder
  Interventions: Other: Text Message; Other: Written reminder
- Plain Text Message (Experimental): plain text message reminder
  Interventions: Other: Text Message; Other: Written reminder
- Written reminder only (Other): written reminder at time of vaccination
  Interventions: Other: Written reminder

INTERVENTIONS:
Other: Text Message
  Arms: Educational Text Message; Plain Text Message
Other: Written reminder

SUMMARY:
Influenza remains a potentially significant and largely preventable source of morbidity and mortality, yet vaccine coverage is low. Young children are at particular risk for underimmunization because they may need to receive 2 doses in a current season. Even among those young children that initiate vaccination, only 40% receive the important second dose, yet one dose does not confer adequate protection. Low-income, urban children may be at particular risk of not receiving two doses. While traditional mail and phone immunization reminders notifying families that a vaccine is due have had limited efficacy in low-income, urban populations, we have demonstrated the success of using text messages. Comparing the effectiveness of different forms of reminders on receipt of this critical second dose of influenza vaccine has not been studied. Besides failure to remember to return for subsequent doses, receipt of 2 doses of influenza vaccine in a season can be affected by limited health literacy regarding influenza vaccination, particularly associated with understanding the need for a second dose since not all children require it. Text messaging offers the ability to combine health literacy promoting information and reminders in a scalable, efficient manner for populations at high risk for underimmunization, limited health literacy, and influenza spread. Therefore, the purpose of this study is to determine whether the provision of interactive vaccine health literacy-promoting information in text message vaccine reminders improves receipt and timeliness of the second dose of influenza vaccine within a season for underserved children in need of two doses.

ELIGIBILITY:
Inclusion Criteria:

* Parenting adult of child age 6 months through 8 years
* Child receives care at study site (visit in last 12 mths)
* child received influenza vaccine and needs a second this season
* Parent has cell phone has text message capability
* Parent speak English or Spanish
* Can read text messages

Exclusion Criteria:

* Parent does not speak English or Spanish
* Parent does not have cell phone with text messages

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Stockwell MS, Hofstetter AM, DuRivage N, Barrett A, Fernandez N, Vargas CY, Camargo S. Text message reminders for second dose of influenza vaccine: a randomized controlled trial. Pediatrics. 2015 Jan;135(1):e83-91. doi: 10.1542/peds.2014-2475. PMID 25548329

RESULTS

PARTICIPANT FLOW:
Groups:
- Educational Text Message: Educational text message reminder
  Text Message
  Written reminder
- Plain Text Message: plain text message reminder
  Text Message
  Written reminder
- Written Reminder Only: written reminder at time of vaccination
  Written reminder
Period: Overall Study
Arm/Group | Educational Text Message | Plain Text Message | Written Reminder Only
Started | 216 | 225 | 219
Completed | 216 | 225 | 219
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Text Message | Plain Text Message | Written Reminder Only | Total
Number analyzed (Participants) | 216 | 225 | 219 | 660
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 216 | 225 | 219 | 660
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 108 | 114 | 327
  Male | 111 | 117 | 105 | 333
Region of Enrollment [Number; unit: participants]
  United States | 216 | 225 | 219 | 660

OUTCOME MEASURES:

1. Primary Outcome: Receipt of 2nd Dose of the Influenza Vaccine.
Time Frame: by April 30th after receipt of first dose (up to 8 months)
Measure: Number; unit: percentage of participants
Arm/Group | Educational Text Message | Plain Text Message | Written Reminder Only
Number analyzed (Participants) | 216 | 225 | 219
percentage of participants | 72.7 | 66.7 | 57.1

2. Secondary Outcome: Number of Subjects Who Receive the 2nd Dose of the Influenza Vaccine on Time.
Time Frame: by 42 days after dose of first vaccination
Population: One patient in the plain text message arm was removed for this analysis because they received the second dose too early and was not re-vaccinated
Measure: Number; unit: percentage of participants
Arm/Group | Educational Text Message | Plain Text Message | Written Reminder Only
Number analyzed (Participants) | 216 | 224 | 219
percentage of participants | 43.5 | 33.9 | 25.6

ADVERSE EVENTS:
Arm/Group | Educational Text Message | Plain Text Message | Written Reminder Only
Serious Adverse Events (participants affected / at risk) | 0/216 | 0/225 | 0/219
Other Adverse Events (participants affected / at risk) | 0/216 | 0/225 | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes